CLINICAL TRIAL: NCT04334876
Title: Rapid SARS-CoV-2 IgG Antibody Testing in High Risk Healthcare Workers and Candidacy for Convalescent Plasma Therapy/Prophylaxis
Brief Title: Rapid SARS-CoV-2 IgG Antibody Testing in High Risk Healthcare Workers
Acronym: COVID-Antibody
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Courtney Rowan, MD, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2003973826
Record Dates: First submitted 2020-04-02; First posted 2020-04-06 (Actual); Results first posted 2021-09-16 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: SARS-CoV-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- High Risk Healthcare Workers (Other): At home, finger prick, antibody test.
  Interventions: Diagnostic Test: SARS-CoV-2 IgG Antibody Testing Kit

INTERVENTIONS:
Diagnostic Test: SARS-CoV-2 IgG Antibody Testing Kit — A, finger prick, at home test for SARS-CoV-2 IgG Antibodies.
  Other Names: Ray Biotech

SUMMARY:
The purpose of this study is to validate the use of a rapid, at home, point-of-care (POC) SARS-CoV-2 IgG antibody test in high risk healthcare workers. Additionally, we would like to evaluate the incidence of seroconversion in this high-risk population and to identify possible candidates for convalescent plasma donation for therapy/prophylaxis.

DETAILED DESCRIPTION:
The success of Singapore, Taiwan and Hong Kong in limiting the impact of the sudden acute respiratory syndrome coronavirus-2 (SARS-CoV-2), also know as COVID-19, has been attributed to their preparedness but mostly to the implementation and distribution of SARS-CoV-2 fast diagnostic tests and establishment of decentralized point-of-care (POC) testing (https://www.nature.com/articles/d41587-020-00010-2). So far, the frontline response to the SARS-CoV-2 outbreak has been polymerase chain reaction (PCR) testing. PCR is the gold standard for diagnosing an infectious agent, and it has the advantage that the primers needed for such tests can be produced with relative speed as soon as the viral sequence is known.

The first quantitative reverse-transcriptase-based PCR (RT-PCR) tests for detecting SARS-CoV2 were designed and distributed in January by the World Health Organization (WHO), soon after the virus was identified. The test protocol is complex and expensive, however, and is mainly suited to large, centralized diagnostic laboratories. Tests typically take 4-6 hours to complete, but the logistical requirement to ship clinical samples means the turnaround time is 24 hours at best. A new fast PCR test (45 min) from Cepheid has been approved by the U.S. Food and Drug Administration on March 21st with availability at the end of the month. Rapid POC tests are also needed to accelerate clinical decision-making and to take some of the workload off centralized test laboratories. Most importantly, the current state of the matter in Indiana University Health system, as well as many around the country is that healthcare workers including from the ER and ICU are currently unable to receive adequate testing through existing facilities. Worst, their access to appropriate personal protective equipment (PPE) has been limited, increasing their exposure risk and causing a significant amount of stress and anxiety for front-line healthcare providers across the country.

Back to the Singapore experience, they have used immunoassays that can provide historic information about viral exposure, as well as diagnostic evidence. They exploited antibody-antigen recognition, either by using monoclonal antibodies (mAbs) to detect viral antigens in clinical samples or by using cloned viral antigens to detect patient antibodies directed against the virus. The lateral flow assay format - essentially a dipstick encased in a cassette - contains the capture reagents (either an mAb directed at a viral antigen or a viral antigen that is recognized by patients' antibodies) immobilized at defined locations on a nitrocellulose membrane, as well as labelled detector mAbs that recognize the same target. A positive result, which is triggered by binding between the analyte and capture mAb and binding by the detector mAb, is visible as a colored line. Two drops of blood from a pinprick is enough to detect a virus. They're essentially the same as home pregnancy kits. Several of these assays are available in Asia, and most European Countries have been using them too. In US, RayBiotech has developed such a similar test using knowledge from the Asian tests (https://www.raybiotech.com/covid-19-igm-igg-rapid-test-kit/). This product is CE marked and certified for diagnostic use in the EU. The application for FDA Emergency Use Authorizations of tests was submitted on March 16th, 2020. At the moment, the FDA has only approved PCR testing. No lateral flow tests have been approved as of March 23rd, 2020. However, this lateral flow test can be used legally in the US, for in vitro diagnostic use, as a POC test when administered by a licensed medical practitioner. These kits were developed in-house by Ray Biotech and validated using samples taken in hospital from patients showing clinical symptoms in Guangzhou China (all confirmed via PCR). Current stocks of 10,000 kits are being replenished daily at RayBiotech, with efforts to increase production ten-fold within the next week. The CE certificate can be found here: https://www.raybiotech.com/files/images/CG-COV_CE-Certificates.jpg.

Based on the Singapore, Taiwan, Hong Kong positive experience, and to curb the fast spread of the virus in the US, we propose to use the POC SARS-CoV-2 IgG Antibody in high risk healthcare workers with or without symptoms, previously quarantine or not. Indeed, we hypothesize that the incidence of seroconversion among ER and ICU healthcare workers is high and higher than current models predict and that several cases are asymptomatic or with mild symptoms.

There are two additional benefits of testing seroconversion.

1. Although there are no official reports, we clearly hear and see selfies of anxiety, stress and exhaustion from our colleagues at the front line. Thus for the healthcare workers knowing that they have seroconverted, will help them be more confident that they are now protected and can work in safer conditions as it has recently been shown that reinfection could not occur in SARS-CoV-2 infected rhesus macaques https://www.biorxiv.org/content/10.1101/2020.03.13.990226v1.
2. The healthcare workers represent an ideal pool of donors for convalescent plasma due to their commitment and the fact that they have usually been tested to give blood or are currently blood donors. The FDA just approved a master protocol for collection and administration of convalescent plasma: https://www.fda.gov/vaccines-blood-biologics/investigational-new-drug-ind-or-device-exemption-ide-process-cber/investigational-covid-19-convalescent-plasma-emergency-inds

In sum, "you cannot fight a fire blindfolded, and we cannot stop this pandemic if we don't know who is infected." (World Health Organization Director-General, 16 March 2020).

If successful and validated, we will hope to rapidly scale it up to propose the rapid SARS-CoV-2 IgG Antibody testing to the general population as has been done in countries that have had almost no death due to COVID-19.

ELIGIBILITY:
Inclusion Criteria:

1. High risk healthcare workers, prioritizing those who are exposed to aerosol generating procedures (physicians and respiratory therapist) working in the emergency room or intensive care units at Indiana University Health or IU school of Medicine affiliated facilities. A second tier of prioritization, to be approached if testing capacity remains after the initial testing phase, will be nurses working these same areas
2. Health care workers who are currently out sick or quarantined due to possible/known exposure to COVID-19 and whose physician confirms that a negative test would allow their return to work are also eligible for testing (Subjects in this group may begin study procedures and be registered once they reach the end of their quarantine period)

Exclusion Criteria:

1. Previously tested for COVID-19

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 571 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2021-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Courtney Rowan, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Health Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Inclusion criteria included High risk healthcare workers, prioritizing those working in the emergency room or intensive care units. A second tier of prioritization, was approached after the initial testing phase, which included expansion to other workers within the healthcare system. We excluded those that had previously tested positive for COVID-19
Period: Overall Study
Arm/Group | High Risk Healthcare Workers
Started | 571
Completed | 500
Not Completed | 71

BASELINE CHARACTERISTICS:
Arm/Group | High Risk Healthcare Workers
Number analyzed (Participants) | 500
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.5 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 388
  Male | 112
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 500
Participant profession [Count of Participants; unit: Participants]
  Physicians | 145
  Nurses | 226
  Respiratory therapist | 33
  other healthcare workers | 95
  Unknown | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participant Health Care Workers With a Positive Rapid, At-home, Point-of-care (POC) SARS-CoV2 IgG Antibody Test.
Description: To determine the number of high risk health care workers with a positive SARS CoV2 IgG on a rapid, at home, self-administered, point-of-care (POC) test. Positive POC tests were then assessed for confirmation using a serum antibody test.
Time Frame: Subjects self-administered the at home POC test and self-reported at their convenience. Testing/reported took approx 15min. Follow up at home testing allowed q 3 weeks post-reporting for a total of 3 at-home tests possible
Population: There was a total of 571 subjects consented. Of these, 71 were lost to follow-up, giving a total of 500 subjects who completed the survey and submitted results for the POC test. Of these 500, 58 subjects did a second follow up point of care test, and 15 patients completed a 3rd test.
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Healthcare Workers
Number analyzed (Participants) | 500
Participants | 8

2. Secondary Outcome: Number of Healthcare Workers Willing to be Convalescent Plasma Donors if Appropriate
Description: To identify possible candidates for convalescent plasma donation for therapy/prophylaxis
Time Frame: Enrollment open from April 2020-January 2021. Subjects completed survey at time of submitting the results of the at home POC test, approximately 15mins.. Survey questioned willingness to donate plasma if found to have antibodies to SARS Co-V2.
Population: We surveyed the number of healthcare workers who would be wiling to donate plasma if found to have positive antibodies to SARS Co-V2 IgG
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Healthcare Workers
Number analyzed (Participants) | 500
Participants | 426

ADVERSE EVENTS:
Time Frame: 6 months
Description: Participants were to report any adverse events to the research team.
Arm/Group | High Risk Healthcare Workers
All-Cause Mortality (participants affected / at risk) | 0/571
Serious Adverse Events (participants affected / at risk) | 0/571
Other Adverse Events (participants affected / at risk) | 0/571

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-26): https://cdn.clinicaltrials.gov/large-docs/76/NCT04334876/Prot_SAP_002.pdf